CLINICAL TRIAL: NCT03679455
Title: A Multicenter, Single-arm, Phase II Study to Evaluate a Safety and Efficacy of Obinutuzumab Induction Followed by 2 Years of Maintenance in Patients With Relapsed/Refractory Waldenström Macroglobulinemia.
Brief Title: A Study of Obinutuzumab (RO5072759) Induction in Patients With Relapsed/ Refractory Waldenström Macroglobulinemia, OBI-1
Acronym: OBI-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Myeloma Consortium (Other)
Collaborators: Roche Pharma AG (Industry); Bioscience, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39235
Record Dates: First submitted 2018-06-04; First posted 2018-09-20 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — obinutuzumab

STUDY DESIGN:
Intervention Model Description: multi-center, single-arm, open label, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Obinutuzumab (RO5072759) 25 MG/ML; Obinutuzumab will be administered by iv. infusion as an absolute (flat) dose of 1000 mg.
  Interventions: Drug: Obinutuzumab 25 MG/ML

INTERVENTIONS:
Drug: Obinutuzumab 25 MG/ML — Study treatment, obinutuzumab is a Type II humanized anti-CD20 monoclonal antibody of the IgG1 subclass derived by humanization of the parental B-Ly1 mouse antibody and produced in the Chinese Hamster Ovary cell line by recombinant DNA technology. The Study Treatment, obinutuzumab is a liquid concentrate for infusion. Obinutuzumab vials are type 1 glass vials with a butyl rubber stopper. Obinutuzumab is provided as a single 1000 mg dose liquid concentrate with a strength of 25 mg/mL. It is supplied in 50 mL glass vials containing 40 mL of the 25 mg/mL liquid concentrate.
  Other Names: Gazyvaro

SUMMARY:
This is a multi-center, single-arm, open label, non-randomized, phase II study designed to investigate the efficacy, safety and tolerability of obinutuzumab given as monotherapy in patients with relapsed/refractory Waldenström Macroglobulinemia (R/R MW).

DETAILED DESCRIPTION:
Study to investigate the efficacy, safety and tolerability of obinutuzumab administered as monotherapy in patients with relapsed/refractory Waldenström Macroglobulinemia (R/R WM)

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to beginning study-related procedures.
2. Male and female subjects aged ≥ 18 years.
3. Able to comply with the study protocol, in the investigator's judgment.
4. Confirmed clinicopathological diagnosis of WM with detectable CD20 positive of the tumor cells
5. Measurable disease defined as serum monoclonal IgM >0.5 g/dL
6. Active disease and indication for treatment based on the Seventh IWWM recommendations (Dimopoulos et al., 2014) defined by presence of at least any one of the following conditions:

   * Recurrent fever, night sweats, weight loss, fatigue
   * Hyperviscosity
   * Lymphadenopathy which is either symptomatic or bulky (≥5 cm in maximum diameter)
   * Symptomatic hepatomegaly and/or splenomegaly
   * Symptomatic organomegaly and/or organ or tissue infiltration
   * Peripheral neuropathy due to WM
   * Symptomatic cryoglobulinemia
   * Cold agglutinin anemia
   * Immune hemolytic anemia and/or thrombocytopenia
   * Nephropathy related to WM
   * Amyloidosis related to WM
   * Hemoglobin ≤10 g/dL
   * Platelet count <100 × 109/L
7. Subjects must have received prior therapies for their WM and have relapsed or refractory WM requiring therapy. Any number of prior therapies is acceptable. Relapsed WM: defined as a subject who has received at least one prior WM therapy and previously achieved a complete or partial remission/response lasting at least 6 months Refractory WM: is defined as progression on treatment; disease progression < 6 months of the last anti-WM therapy
8. Subjects must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count ≥ 1.5 x 109/l (unless decreased due to WM involvement of the bone marrow)
   * Platelets ≥ 75 x 109/l (unless decreased due to WM involvement of the bone marrow)
   * Hemoglobin ≥ 9 g/dL
   * Total bilirubin ≤ 1.5 x ULN or < 2 x ULN if attributable to hepatic infiltration by neoplastic disease
   * AST and ALT < 2.5 x ULN
   * Calculated creatinine clearance by Cockcroft-Gault formula >40 mL/min
   * INR ≤ 1.5
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
10. Fertile men or women of childbearing potential, unless ≥ 2 years after the onset of menopause (for women), must be willing to use a highly effective contraceptive method (Pearl Index < 1) such as oral contraceptives, intrauterine device, sexual abstinence or barrier method of contraception in conjunction with spermicidal jelly, during study treatment and for 18 months after end of obinutuzumab treatment.

Exclusion Criteria:

1. Lactating women, women with a positive pregnancy test at Visit 1 or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through 18 months after end of obinutuzumab treatment.
2. Known involvement of the central nervous system by WM.
3. Vaccination with a live vaccine a minimum of 28 days prior to study enrolment (vaccination day considered as Day 0).
4. History of stroke or intracranial hemorrhage within 12 months prior to study enrollment.
5. Currently active, clinically significant cardiovascular disease.
6. Any active systemic infection. Caution should be exercised when considering the use of obinutuzumab in patients with a history of recurring or chronic infections.
7. Positive for hepatitis C antibody at screening.
8. Positive test result for chronic hepatitis B virus (HBV) infection (defined as a positive HBsAg serology). Patients with occult or prior HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive total hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing during treatment and follow-up until 12 months after the last dose of obinutuzumab.
9. Known HIV infection at screening.
10. Any serious illness, medical condition, organ system dysfunction or abnormality in clinical laboratory test that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
11. Concurrent use of other anti-cancer agents or treatments.
12. Prior use of any investigational monoclonal antibody therapy within 6 months of study start.
13. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy, known hypersensitivity to any of the study drugs or sensitivity to murine products.
14. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives or 4 Weeks prior to first study treatment dose, whichever is longer, or participation in any other interventional clinical study.
15. Prior use of radiation therapy within 4 weeks of enrollment.
16. History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
17. History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response (BOR) | Up to 3,5 years
  BOR is the best response recorded from the start of the treatment until disease progression: response assessments recorded as CR, VGPR, PR, MR, SD, PD. As a responder is considered patient with at least MR (CR, VGPR, PR, MR). BOR will be presented as rates with corresponding exact 95% CI.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3,5 years
  PFS will be calculated as time from fist treatment dose until progression or death of any cause. The PFS will be defined as well-documented and verifiable data. The Kaplan-Meier curve will be provided. The median time to PFS along with associated 95% confidence interval will be provided as well.
Overall Survival (OS) | from first study treatment dose till 1 year after the treatment period
  OS is defined as time from first study treatment dose to death due to any cause. Survival distributions will be estimated using the Kaplan-Meier method. Each subject will be followed for 1 year after the treatment period.
Overall Response Rate (ORR) | after 6 Cycles of obinutuzumab treatment (after induction phase); each cycle is 21 days in Induction Phase;
  ORR as a secondary endpoint will be assessed after completion of induction phase and after maintenance phase. Responders include subjects with at least MR (CR, VGPR, PR, MR). Non-responders include subjects with Stable Disease (SD) and Progressive Disease (PD). Subjects with unknown or missing responses will be considered as non-responders.
Overall Response Rate (ORR) | after all 12 Cycles of treatment in Maintenance Phase (at first visit in follow-up phase FU2M) or after the last dose, if not after 12 Cycles of obinutuzumab (each cycle is 8 weeks in Maintenance Phase;
  ORR as a secondary endpoint will be assessed after completion of induction phase and after maintenance phase. Responders include subjects with at least MR (CR, VGPR, PR, MR). Non-responders include subjects with Stable Disease (SD) and Progressive Disease (PD). Subjects with unknown or missing responses will be considered as non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Wróbel, MD.PhD, Principal Investigator — USK Wrocław
Locations (2):
- Poland (2):
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu; Oddział Hematologii i Transplantacji Szpiku, Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital kliniczy im. Jana Mikulicza-Radeckiego we Wrocławiu; Klinika Hematologii, Nowotworów Krwi Transplantacji Szpiku, Wroclaw, Lower Silesian Voivodeship

REFERENCES:
- [Derived] Wrobel T, Kalicinska E, Zaucha JM, Morawska M, Giannopoulos K, Jamroziak K, Lech-Maranda E, Taszner M, Szeremet A, Malecki B, Druzd-Sitek A, Lojko-Dankowska A, Dytfeld D. Obinutuzumab induction and maintenance in patients with Waldenstrom macroglobulinaemia: an open-label, single-arm phase 2 study. EClinicalMedicine. 2025 Jul 25;86:103383. doi: 10.1016/j.eclinm.2025.103383. eCollection 2025 Aug. PMID 40756965